CLINICAL TRIAL: NCT01967849
Title: Prevalence of Carbohydrate Intolerance in Lean and Overweight/Obese Children
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 9909011190; R01HD040787 (NIH); 1R01DK111038-01A1 (NIH); 2R01HD028016-20A1 (NIH)
Record Dates: First submitted 2013-07-15; First posted 2013-10-23 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Obesity; Type 2 Diabetes
Keywords: obesity; type 2 diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA blood sample is obtained from IV during oral glucose tolerance test.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Obese/overweight chldren/adolescents: Obese or overweight children and adolescents between ages 7-21 that are at risk for developing type 2 diabetes will undergo an Oral Glucose Tolerance test (OGTT) to asses glucose status.
  Interventions: Diagnostic Test: Oral Glucose tolerance test
- Lean children/adolescents: Lean children/adolescents between the ages of 7-21. This cohort should have family members that have type 2 diabetes or was the result of a gestational diabetes pregnancy. They will undergo an Oral Glucose Tolerance Test to assess glucose status.
  Interventions: Diagnostic Test: Oral Glucose tolerance test

INTERVENTIONS:
Diagnostic Test: Oral Glucose tolerance test

SUMMARY:
The purpose of this study is to determine the prevalence of impaired glucose (carbohydrate) tolerance in lean children with a family history of diabetes and in overweight/obese children with or without a family history of diabetes mellitus.

DETAILED DESCRIPTION:
The patient participates in the study for a total duration of approximately four hours. The study nurse will do a nursing assessment, including measuring the patient's height, weight, waist circumference, hip circumference, blood pressure, and pulse, along with evaluation of acanthosis nigricans and striae rubrae. The patient's percent body fat, fat mass and lean mass may also be measured using a Tanita scale. The nurse will obtain a family and medical history from the patient and/or the patient's parent/guardian. In addition, before starting the oral glucose tolerance test (OGTT), the nurse will request a urine sample from the patient for analysis of microalbumin and creatinine.

The patient will receive 1.75 g/kg to a maximum of 75 g of a sugar drink, orally (Glucola). The patient will have one intravenous line. "Emla" or a local anesthetic (0.1cc buffered lidocaine) will be applied before the placement of the IV catheter. Blood will be drawn 10 times over three hours. Should abnormal glucose results be found, appropriate referrals will be made. We will draw approximately 80 cc of blood during this study. The blood will be analyzed for glucose, lactate, insulin, proinsulin, c-peptide, interleukin-6, tumor necrosis factor-α(TNF), free fatty acids (FFAs), enhanced lipid profile, leptin, and adiponectin as well as an optional 10 cc sample to be stored for future undetermined analysis.

ELIGIBILITY:
Inclusion Criteria:

* ages 7-21
* family history of type 2 diabetes mellitus

Exclusion Criteria:

* Children will be excluded if they have previously been treated for another endocrinopathy or are on any chronic medications that are known to alter glucose or insulin metabolism, such as oral steroids, or certain psychiatric medications, such as Xeleca, Lithium and Paxil.
* Lean (not overweight or obese) will be defined as a body mass index (BMI) (kg/m2) less than the 85th percentile specific for age and gender, overweight will be defined as a BMI between the 85th and 95th percentiles, and obesity will be defined as a BMI greater than the 95th percentile.
* Children will be excluded from participating in the genetic analysis if they are treated oral glucocorticoids or antirejection or chemotherapy (e.g. tacrolimus, Lasparaginase.

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Primarily these patients are recruited from Yale Pediatric Endocrinology Clinic or are siblings of patients.
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 1999-09 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2023-09-18 (Actual)

PRIMARY OUTCOMES:
Glucose Tolerance | Baseline measurements
  Glucose tolerance status as determined by 3 hour oral glucose tolerance test

SECONDARY OUTCOMES:
Insulin resistance | Completed at baseline measurement
  Insulin secretion measured during OGTT by variety of insulin resistance calculations (WBISI, DI, IGI, HOMA-IR)

OTHER OUTCOMES:
Gene Expression | Completed at baseline measurement
  Gene mutation/allelle variation identification measured via gene extraction

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Caprio, MD, Principal Investigator — Yale Pediatric Endocrinology
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trico D, McCollum S, Samuels S, Santoro N, Galderisi A, Groop L, Caprio S, Shabanova V. Mechanistic Insights Into the Heterogeneity of Glucose Response Classes in Youths With Obesity: A Latent Class Trajectory Approach. Diabetes Care. 2022 Aug 1;45(8):1841-1851. doi: 10.2337/dc22-0110. PMID 35766976
- [Derived] Halloun R, Galderisi A, Caprio S, Weiss R. Lack of Evidence for a Causal Role of Hyperinsulinemia in the Progression of Obesity in Children and Adolescents: A Longitudinal Study. Diabetes Care. 2022 Jun 2;45(6):1400-1407. doi: 10.2337/dc21-2210. PMID 35235641
- [Derived] Zabarsky G, Beek C, Hagman E, Pierpont B, Caprio S, Weiss R. Impact of Severe Obesity on Cardiovascular Risk Factors in Youth. J Pediatr. 2018 Jan;192:105-114. doi: 10.1016/j.jpeds.2017.09.066. PMID 29246331
- [Derived] Hershkop K, Besor O, Santoro N, Pierpont B, Caprio S, Weiss R. Adipose Insulin Resistance in Obese Adolescents Across the Spectrum of Glucose Tolerance. J Clin Endocrinol Metab. 2016 Jun;101(6):2423-31. doi: 10.1210/jc.2016-1376. Epub 2016 Apr 7. PMID 27054297